CLINICAL TRIAL: NCT06192342
Title: Baseline Ventilatory Parameters in Patients With Acute Neurological Injury
Brief Title: Ventilatory Parameters in Acute Neurological Injury
Status: Recruiting | Type: Observational
Sponsor: Ramos Mejía Hospital (Other)
Responsible Party: Principal Investigator, Roberto Santa Cruz, Principal Investigator, Ramos Mejía Hospital
Other Study IDs: Observational
Record Dates: First submitted 2023-12-04; First posted 2024-01-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-06

CONDITIONS: Neurologic Decompensation, Acute; Traumatic Brain Injury; Stroke; Subarachnoid Hemorrhage
Keywords: acute neurological injury, mechanical ventilation
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute neurological injury: Patients ≥ 16 years of age with ANI requiring mechanical ventilation for neurological causes, without baseline lung injury, defined by a PaO2/FiO2 ≥ 300 and with a normal chest x-ray

SUMMARY:
The goal of this observational study is to test the association between baseline ventilatory parameters (in particular mechanical power (MP), mechanical power normalized to predicted body weight (MP/PBW) and driving pressure (DP) with the baseline neurological status (assessed through the Glasgow coma score) in adults patients under mechanical ventilation with acute neurological injury secondary to stroke, brain trauma or subarachnoid hemorrhage.

The main question[s]it aims to answer are:

1. In patients with acute neurological injury under mechanical ventilation, is there a correlation between the acute neurological injury, assessed using the Glasgow scale on admission, and baseline ventilatory parameters?
2. In patients with acute neurological injury under mechanical ventilation, are the baseline ventilatory parameters altered at baseline?

DETAILED DESCRIPTION:
Adults patients with acute neurological injury (ANI) secondary to stroke, brain trauma or subarachnoid hemorrhage may present extraneurological complications. They occur as a consequence of the release of inflammatory mediators in an altered blood-brain barrier, which reach the circulation and thus alter the functionality of other organs. Of the affected organs, the lung is the most frequently compromised, leading to increased morbidity, mortality, and worse neurological outcomes. It should be noted that a large proportion of patients with ANI require mechanical ventilation (MV), which also through the production of inflammatory mediators, can lead to the development of ventilator-induced lung injury (VILI) and alteration of other organs.

From the above, it can be thought that in patients with ANI, the basal respiratory parameters could be altered and this is important, given that in this group of patients, the ventilatory parameters could generate changes at the brain level, particularly an increase in intracranial pressure (ICP) and variation in PaCO2 that would produce changes in the vasculature and concomitantly in cerebral blood flow. In turn, the use of protective ventilation, recommended in other pathologies such as acute respiratory distress syndrome (ARDS), is not clearly defined for this group of patients. For this reason, the objective of this study is the assessment of baseline ventilatory parameters in patients with ANI, in particular mechanical power (MP), mechanical power normalized to predicted body weight (MP/PBW) and driving pressure (DP) and to determine their association with the baseline neurological status (assessed through the Glasgow coma score). The hypothesis of the study, assuming that the greater the initial neurological damage, the greater the ventilatory alterations, is that MP correlates with the degree of neurological injury. The second hypothesis is that ventilatory variables, particularly MP, are altered at baseline in patients with LNA.

ELIGIBILITY:
Inclusion Criteria:

Acute neurological injury in patients ≥ 16 years of age with requiring mechanical ventilation for neurological causes and without baseline lung injury, defined as: normal chest x-ray and adequate oxygenation; PaO2/FiO2 ≥ 300.Neumovent TS and Neumovent Advance respirators will be used.

-

Exclusion Criteria:

Pneumothorax, or a pleural drainage tube. Hemodynamic instability (mean blood pressure ≤ 65 mmHg) or high doses of inotropes (Norepinephrine > 0.5 gammas/kilo/minute or equivalent).

PaO2/FiO2 < 80 mmHg. Chronic obstructive pulmonary disease (COPD). Pregnant

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients ≥ 16 years of age with an ANI requiring mechanical ventilation for neurological causes.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between acute neurological injury and mechanical power normalized to predicted body weight | The first 2 days of the patient on mechanical ventilation (MV)
  To determine the degree of correlation between acute neurological injury, assessed using the Glasgow coma score [GCS; with a score between 3 (worst score, most severe) and 15 (best score, least severe)] and mechanical power normalized to predicted body weight (Joules/minute/kilograms)

SECONDARY OUTCOMES:
Correlation between acute neurological injury and mechanical power | The first 2 days of the patient on mechanical ventilation (MV)
  To determine the degree of correlation between acute neurological injury, assessed using the Glasgow coma score [GCS; with a score between 3 (worst score, most severe) and 15 (best score, least severe)] and mechanical power (Joules/minute)
Correlation between acute neurological injury and ΔP | The first 2 days of the patient on mechanical ventilation (MV)
  To determine the degree of correlation between acute neurological injury, assessed using the Glasgow coma score [GCS; with a score between 3 (worst score, most severe) and 15 (best score, least severe)] and ΔP (centimeter of water)
To assess static pressure | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the static pressure: Pplat (centimeter of water)
To assess the respiratory system resistance | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the respiratory system resistance: it is the relationship between the difference between peak pressure and static pressure with the inspiratory flow: R = (Ppeak-Pplat)/Inspiratory flow (centimeter of water/liters/second)
To assess the driving pressure | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the driving pressure: it is the difference between static pressure and PEEP: ΔP = Pplat-PEEP (centimeter of water)
To assess the static compliance | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the static compliance: it is the relationship between tidal volume and ΔP (mililiters/centimeter of water)
To assess the dynamic driving pressure | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the dynamic driving pressure: it is the difference between peak pressure and PEEP: ΔP = Ppeak-PEEP (centimeter of water), (centimeter of water)
To assess mechanical power normalized to predicted body weight | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the mechanical power normalized to predicted body weight (Joules/minute/kilograms)
To assess the static pressure according to the different subgroups of ANI | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the static pressure (centimeter of water) according to the different subgroups of ANI: brain trauma injury (BTI), subarachnoid hemorrhage (SAH) and stroke.
To assess the respiratory system resistance according to the different subgroups of ANI | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the respiratory system resistance (it is the relationship between the difference between peak pressure and static pressure with the inspiratory flow) (centimeter of water/liters/seconds), according to the different subgroups of ANI: brain trauma injury (BTI), subarachnoid hemorrhage (SAH) and stroke.
To assess the driving pressure according to the different subgroups of ANI | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the driving pressure (it is the difference between static pressure and PEEP) (centimeter of water), according to the different subgroups of ANI: brain trauma injury (BTI), subarachnoid hemorrhage (SAH) and stroke.
To assess the static compliance according to the different subgroups of ANI | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the static compliance (it is the relationship between tidal volume and ΔP) (mililiters/centimeter of water), according to the different subgroups of ANI: brain trauma injury (BTI), subarachnoid hemorrhage (SAH) and stroke.
To assess the dynamic driving pressure according to the different subgroups of ANI | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the dynamic driving pressure (it is the difference between peak pressure and PEEP) (centimeter of water), according to the different subgroups of ANI: brain trauma injury (BTI), subarachnoid hemorrhage (SAH) and stroke.
To assess the mechanical power normalized to predicted body weight according to the different subgroups of ANI | The first 2 days of the patient on mechanical ventilation (MV)
  To assess the mechanical power normalized to predicted body weight (Joules/minute/kilograms) according to the different subgroups of ANI: brain trauma injury (BTI), subarachnoid hemorrhage (SAH) and stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Santa Cruz, Principal Investigator — Hospital General Ramos Mejia
Locations (1):
- Roberto Santa Cruz, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina